CLINICAL TRIAL: NCT00839605
Title: Dexmedetomidine and Hypoxic Pulmonary Vasoconstriction in Thoracic Surgical Procedure and One-Lung Ventilation(OLV)
Brief Title: Dexmedetomidine and Hypoxic Pulmonary Vasoconstriction in Thoracic Surgical Procedures and One-Lung Ventilation
Acronym: Dex-One-Lung
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 1124100 Hospira
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Cancer; Lung Cancer; Chest Wall Disorders
Keywords: Thoracic surgery one lung ventilation; airway reconstruction
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dexmedetomidine: Those requiring thoracic surgery and receiving dex
  Interventions: Drug: Dexmedetomidine
- placebo: Group having thoracic surgery and not receiving dex drug

INTERVENTIONS:
Drug: Dexmedetomidine — loading dose:0.3mcg/kg. Infusion of 0.3mcg/kg/hr
  Other Names: Precedex
  Groups: Dexmedetomidine

SUMMARY:
The purpose of this study is to evaluate the effects of Dexmedetomidine when used during thoracic surgery.

The primary outcome will be changes in oxygenation as measured the PaO2 during one lung ventilation.

DETAILED DESCRIPTION:
To collect data on the effects of Dexmedetomidine(DEX)(0.3mcg/kg loading dose followed by an infusion of 0.3mcg/kg/hr)on Hypoxic pulmonary vasoconstriction when administered to patients during surgery with one lung ventilated thoracic procedures. Dexmedetomidine has both vasoconstricting and vasodilatatory effect on peripheral vasculature but its effect on pulmonary vessels is not known. If it is predominantly a vasodilator on pulmonary vessels it can inhibit hypoxic pulmonary vasoconstriction and will increase shunting of venous blood to arterial circulation without oxygenation. If our study proves it to be a vasodilator for pulmonary vessels then it will not be wise to use it in thoracic procedure with one lung ventilation. If our study proves that it is a vasoconstrictor for pulmonary vessels, then it will be an excellent adjunct to other anesthetic agents during one lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age.
2. Subject is American Society of Anesthesiologists (ASA) Physical Status I, II, III, or IV.
3. If female, subject is non-lactating and is either:

   * Not of childbearing potential, defined as post-menopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
   * Of childbearing potential but is not pregnant at time of baseline and is practicing one of the following methods of birth control: oral or parenteral contraceptives, double-barrier method, vasectomized partner, or abstinence from sexual intercourse.
4. Subject requires thoracic surgical procedure .
5. Subject (or subject's legally authorized representative) has voluntarily signed and dated the informed consent document approved by the Institutional Review Board.

Exclusion Criteria:

1. Subject has received general anesthesia within 7 days prior to study entry, has received any experimental drug within 30 days prior to study drug administration, or has been previously enrolled in this study.
2. Subject has central nervous system (CNS) disease with an anticipated potential for increased intracranial pressure, an uncontrolled seizure disorder and/or known psychiatric illness that could confound a normal response to sedative treatment.
3. Subject has received treatment with an alpha-2 agonist or antagonist within 14 days of the scheduled surgery/procedure.
4. Subject for whom opiates, benzodiazepines, DEX or other alpha-2 agonists are contraindicated.
5. Subject has received an IV opioid within one hour, or PO/IM opioid within four hours, of the start of study drug administration.
6. Subject has acute unstable angina, acute myocardial infarction documented by laboratory findings in the past six weeks, heart rate < 50 bpm, SBP < 90 mmHg, or third-degree heart block unless patient has a pacemaker.
7. Subject has known elevated SGPT (ALT) and/or SGOT (AST) values of > 2 times the upper limit of normal (ULN) within the two months prior to screening, and/or a history of liver failure.
8. Subject has any other condition or factor which, in the Investigator's opinion, might increase the risk to the subject.
9. On vasodilators, i.e.,nitroglycerin, nitroprusside, or ACE inhibitors
10. on vasopressors, i.e, norepinephrine,epinephrine, or vasopressin

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients whom will be receiving thoracic surgery
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be changes in oxygenation measured by the PaO2 during one lung ventilation | During thoracic surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: joseph tobias, md, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No